CLINICAL TRIAL: NCT06097806
Title: Effects of Different Fresh Gas Flows on Carboxyhemoglobin Levels
Brief Title: Effects of Different Fresh Gas Flows on Carboxyhemoglobin Levels and Postoperative Patient Outcomes in Pediatric Cardiovascular Surgery
Status: Recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Selin Saglam, Specialist, Başakşehir Çam & Sakura City Hospital
Other Study IDs: Başakşehir Çam and Sakura
Record Dates: First submitted 2023-10-06; First posted 2023-10-24 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Low Flow Anesthesia; High Flow Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low-flow anesthesia group: In this group, ventilation parameters is adjusted to have fresh gas flow/minute ventilation ratio below 0.5
  Interventions: Other: low and high flow
- High-flow anesthesia group: In this group, ventilation parameters is adjusted to have fresh gas flow/minute ventilation ratio above 1.0
  Interventions: Other: low and high flow

INTERVENTIONS:
Other: low and high flow — low and high flow anesthesia are both being used. The effects of different gas flows will be evaluated.

SUMMARY:
Low flow anesthesia; It is an anesthesia practice in which, after absorbing at least 50% of the exhaled air and carbon dioxide (CO2) using a semi-closed rebreathing system, the unused anesthetic gases are mixed with a certain amount of fresh gas and then completely or partially returned to the patient in the next inspiration. Theoretically, when low flow anesthesia is compared to high or normal flow anesthesia; it is known to have advantages such as using less inhalation agent, preserving mucociliary activity, preventing microatelectasis, preserving the amount of moisture, and reducing temperature loss.

In studies conducted in different fresh gas flows, it has been observed that CO, which is thought to accumulate in the body by rebreathing in a closed circuit, increases as a result of the chemical interaction and dry CO2 absorbent. However, there is no evidence in these studies that low-flow anesthesia increases CO accumulation and alters hemodynamics.

In our clinic, low-flow and high-flow anesthesia technics are both being used. In this study, we aimed to evaluate the effects of high- and low-flow sevoflurane anesthesia applied with a closed system on perioperative carboxyhemoglobin (COHb) levels and hemodynamic system in pediatric cardiovascular surgery cases.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 2 months and 7 years undergoing elective cardiac surgery
* American Society of Anesthesiology (ASA) score II ve III patients

Exclusion Criteria:

* Patients undergoing emergency surgery
* Patients who need mechanical ventilation or any respiratory support before the operation
* Patients with left to right shunt
* cyanotic patients
* Patients younger than 2 months and older than 7 years

Ages: 2 Months to 7 Years | Sex: All
Age Groups: Child
Study Population: Patients will be selected among the patients who will undergo cardiac surgery at Basaksehir Cam and Sakura City Hospital Pediatric Cardiovascular Surgery Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
COHb levels | at the 30th minute of the surgery, at the beginning of cardiopulmonary bypass, at the time of chest closure, at the time of intensive care unit admission
  COHb values will be measured in arterial blood gas samples at different fresh gas flow levels.

SECONDARY OUTCOMES:
extubation time | at the time that patient is extubated up to 24 hours
  the time of extubation
body temperature | at the 30th minute of the surgery, at the beginning of cardiopulmonary bypass, at the time of chest closure, at the time of intensive care unit admission
  body temperature
bleeding | 24 hours
  Total amount of bleeding during the first 24 hours
vasoactive inotrope score (VIS) | postoperative first hour
  VIS at the end of the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)